CLINICAL TRIAL: NCT06956365
Title: Van Yuzuncu Yil University Faculty of Medicine Ethics Committee
Brief Title: To Compare the Effects of Oxytocin and Carbetocin on Intraoperative Hemodynamic Changes in Cesarean Section Surgeries.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Nurettin KURT, Assistant Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/09-10
Record Dates: First submitted 2023-08-22; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Cesarean Section
Keywords: Cesarean section; Oxytocin; Carbetocin; Uterotonic; Intraoperative bleeding
MeSH Terms: conditions — Blood Loss, Surgical | interventions — O-antigen, Acinetobacter strain 90

STUDY DESIGN:
Intervention Model Description: In 80 pregnant patients scheduled for elective cesarean section, patients will be randomly assigned to receive 5 IU oxytocin or 100 μg carbetocin IV bolus intraoperatively after the birth of the baby.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Group-O) (Active Comparator): Group-O: Oxytocin group (n:40). In cesarean surgery, 5 IU of oxytocin will be administered after the baby delivered.
  Interventions: Procedure: Group-O
- Carbetocin (Group-C) (Experimental): Group-C: Carbetocin group (n:40). In cesarean surgery, 100 μg carbetocin IV bolus will be administered after the baby delivered.
  Interventions: Procedure: Group-C

INTERVENTIONS:
Procedure: Group-C — 100 iu carbetosin administered to carbetocin group
  Other Names: Group Carbetosin
  Arms: Carbetocin (Group-C)
Procedure: Group-O — In cesarean surgery, 5 IU of oxytocin will be administered after the baby delivered.
  Other Names: Group Oxytocine
  Arms: Oxytocin (Group-O)

SUMMARY:
To compare the effects of oxytocin and carbetocin, used as uterotonics in elective caesarean section surgeries, in terms of intraoperative hemodynamic changes.

DETAILED DESCRIPTION:
The study will have a double-blind design and will be conducted after obtaining an approval from the local ethics committee. The study will include 80 patients planned for elective caesarean section surgeries , aged 18-40 years with an ASA score of I-II. The patients will be randomized by sealed tender and will be divided into 2 groups with 40 patients each.

All cases will receive routine preparation for general anesthesia. All patients placed on the operating room will receive two large-bore vascular access. For anesthesia induction 2 mg/kg propofol and 0.5 mg/kg rocuronium will be used. Anesthesia will be maintained with 60% air, 40% oxygen and 2 MAC sevoflurane.Demographic data of the patients (age, height, weight), ASA score and surgical time will be recorded. During the operation, hemodynamic parameters will be recorded just before the drugs are given and at the 1st, 5th, 10th, 15th, 20th, 25th and 30th minutes after the drug is given. In addition, intraoperative blood loss and the need for additional uterotonics throughout the surgery will be recorded. All data will be recorded and statistical analysis will be made.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for caesarean sections
* Between 18-40 years
* ASA I-II group
* Those who will undergo general anesthesia
* Those between 35-40 weeks of pregnancy
* 1st and 2nd caesarean sections

Exclusion Criteria:

* Those who prefer spinal or epidural anesthesia
* Those who are outside the age range of 18-40
* Those who are ASA III and above
* Those with HT, DM, cardiac and respiratory diseases
* Preeclampsia, eclampsia, HELLP
* Those with a history of drug use that affects the cardiovascular system
* Placenta Previa, Placenta Acreta, Placenta Acreta

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Uterine tonus | For 30 minutes after carbetocin administration.
  The effect of carbetocin on uterine tone will be evaluated by the surgical team using a numerical scoring scale between 0-10. A score of 0 will indicate atony, and a score of 10 will indicate full contraction.
Additional uterotonic drug requirement | For 30 minutes after carbetocin administration.
  If the uterine tone is 7 or below, the surgical team will perform uterine massage, and in patients who do not see a sufficient increase in uterine tone, an additional uterotonic, 0.2 mg methylergonavine (Methyl ampoule 0.2 mg/ml) will be administered IM by the anesthesia team and recorded.

SECONDARY OUTCOMES:
Intraoperative bleeding | from drug administration to the end of surgery.
  Total intraoperative bleeding was recorded by calculating and estimating the aspirator volume, pad-sponge-compress count and surgical area.
Mean Blood Pressure | Intraoperatively every 5 minutes
  Mean blood pressure will be measured every 5 minutes intraoperatively using a noninvasive method.
Heart Rate | Intraoperatively every 5 minutes
  Heart rate will be measured every 5 minutes intraoperatively using a noninvasive method.

CONTACTS AND LOCATIONS:
Overall Officials: Şükran ŞS Sevimli, Assoc.Prof, Study Director — Van Yüzüncü Yıl University Van/Turkey
Locations (1):
- Van Yuzuncu Yil University, Van, Tuşba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study protocol anda statistical analysis plan will be share with other researchers
Supporting Information: Study Protocol, SAP
Time Frame: 10 months
Access Criteria: The access can be provided via the e-mail addresses below dr.nurettinkurt@gmail.com

REFERENCES:
- [Background] He G, Li LI, Guan E, Chen J, Qin YI, Xie Y. Fentanyl inhibits the progression of human gastric carcinoma MGC-803 cells by modulating NF-kappaB-dependent gene expression in vivo. Oncol Lett. 2016 Jul;12(1):563-571. doi: 10.3892/ol.2016.4619. Epub 2016 May 25. PMID 27347181
- [Background] Dutriez-Casteloot I, Emmanuelli V, Wiart JF, Tavernier A, Besengez C, Storme L, Houfflin-Debarge V. Long-Lasting Analgesia With Transdermal Fentanyl: A New Approach in Rat Neonatal Research. Front Pharmacol. 2022 Mar 17;13:798011. doi: 10.3389/fphar.2022.798011. eCollection 2022. PMID 35370716
- [Background] Clemensen J, Rasmussen LV, Abelson KSP. Transdermal Fentanyl Solution Provides Long-term Analgesia in the Hind-paw Incisional Model of Postoperative Pain in Male Rats. In Vivo. 2018 Jul-Aug;32(4):713-719. doi: 10.21873/invivo.11299. PMID 29936450